CLINICAL TRIAL: NCT00735046
Title: Cognitive Behavioural Resource-based Therapy of Early Dementia in the Everyday Setting
Brief Title: Cognitive Behavioural Therapy of Early Dementia
Acronym: KORDIAL
Status: Completed | Type: Observational
Sponsor: Technical University of Munich (Other)
Collaborators: University of Leipzig (Other); Zentralinstitut für Seelische Gesundheit Mannheim (Other); Humboldt-Universität zu Berlin (Other)
Responsible Party: Alexander Kurz M.D., klinikum rechts der Isar
Other Study IDs: KOR-683-KUR-0000-I
Record Dates: First submitted 2008-08-13; First posted 2008-08-14 (Estimated); Last update posted 2011-01-14 (Estimated); Status verified 2008-07

CONDITIONS: Dementia
Keywords: Early dementia in Alzheimer's disease (MMSE ≥ 21)
MeSH Terms: conditions — Dementia | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: None Retained — not required
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Intervention
  Interventions: Behavioral: Cognitive behavioral therapy for early Alzheimer's disease
- 2: control
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy for early Alzheimer's disease — 12 weekly individual sessions, total duration 3 months, regular involvement of patient's proxy ever second session. Intervention is manualized but is flexible with regard to individual resources and needs.
  Groups: 1
Other: Control — Patients and proxies who are assigned to treatment as usual
  Groups: 2

SUMMARY:
A randomized, controlled, parallel-group trial to evaluate the efficacy of a cognitive behavioral therapy for patients with early dementia.

DETAILED DESCRIPTION:
The KORDIAL study is a randomized, controlled, parallel-group trial evaluating the efficacy of a cognitive behavioral therapy for patients at the early stage of Alzheimer's disease. The 3-month experimental intervention consists of 12 individual sessions with regular involvement of carers or other patient proxies. Strategies for improving the patient's coping ability and for enhancing their psychological well-being are combined. The primary outcome criterion is functioning in the everyday context after completion of the intervention and after another 6 months. The control condition will be treatment as usual. The study will be conducted in 5 university outpatient units and in 5 specialist offices.

ELIGIBILITY:
Inclusion Criteria:

* Mild dementia (MMSE > 21) in Alzheimer's disease (ICD-10), proxy available

Exclusion Criteria:

* Acute of unstable psychiatric or physical disease, proxy unavailable
* Participation in another trial

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to memory clinics and specialist (psychiatrist, neurologist) offices
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2008-04; Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Functional ability in the everyday context | Baseline, post treatment, 6 months post treatment

SECONDARY OUTCOMES:
Quality of life, depression, neuro-psychiatric symptoms | Same as for primary outcome

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Kurz, MD, Study Director — Klinikum rechts der Isar
Locations (1):
- Prof. Dr. A. Kurz, Department of Psychiatry and Psychotherapy, Klinikum rechts der Isar, Technische Universitaet Muenchen, Munich, Bavaria, Germany

REFERENCES:
- [Background] Kliegel M, Eschen A, Thone-Otto AI. Planning and realization of complex intentions in traumatic brain injury and normal aging. Brain Cogn. 2004 Oct;56(1):43-54. doi: 10.1016/j.bandc.2004.05.005. PMID 15380875
- [Background] Werheid K, Thone-Otto AI. [Cognitive training in Alzheimer's dementia]. Nervenarzt. 2006 May;77(5):549-57. doi: 10.1007/s00115-005-1998-2. German. PMID 16228161
- [Background] Kurz A, Pohl C, Ramsenthaler M, Sorg C. Cognitive rehabilitation in patients with mild cognitive impairment. Int J Geriatr Psychiatry. 2009 Feb;24(2):163-8. doi: 10.1002/gps.2086. PMID 18636436